CLINICAL TRIAL: NCT03583632
Title: Visual Acuity and Optical Coherence Tomography One Year After Peeling of Epiretinal Membranes
Status: Completed | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of the Department of Ophthalmology, Professor, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: ERM 1year follow-up
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: visual acuity testing — testing of visual ycuity by ETDRS charts
Device: optical coherence tomography — optical coherence tomography generates sectional slides of the retinal tomography with light

SUMMARY:
Improvement in visual acuity and retinal anatomy one year after surgery is assessed and compared to data preoperative and 3 months after surgery

DETAILED DESCRIPTION:
Improvement in visual acuity and retinal anatomy (documented by optical coherence tomography) one year after surgery is assessed and compared to data preoperative and 3 months after surgery. Improvements in retinal morphology are analysed by remission of optical coherence biomarkers after surgery. Aim of the study is to examine possible improvements of surgical outcomes in the period up to the one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* vitrectomy with Membrane Peeling due to an epiretinal membrane

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: For this study only patients after vitrectomy with Membrane Peeling due to epiretinal membranes are selected
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
visual acuity | 3 minutes
  visual acuity testing with EDTRS charts

SECONDARY OUTCOMES:
optical coherence tomography | 3 minutes
  optical coherence tomography generates slides of the retinal anatomy with light

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Prof, Principal Investigator — VIROS at Hanuschkrankenhaus Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria